CLINICAL TRIAL: NCT01160341
Title: Phase 4 Study of About the Effect of Testosterone Treatment on the Components of Metabolic Syndrome
Brief Title: Metabolic Syndrome Criteria and the Effect of Testosterone Treatment in Young Men With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Dr. Alper Sonmez, Gulhane School of Medicine Department of Endocrinology and Metabolism
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GSM-072010
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-01

CONDITIONS: Hypogonadism
Keywords: Metabolic syndrome; Hypogonadism; Testosterone
MeSH Terms: conditions — Hypogonadism; Metabolic Syndrome | interventions — Testosterone Propionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosteron, secondary hypogonadism (Experimental)
  Interventions: Drug: Testosteron

INTERVENTIONS:
Drug: Testosteron — Testosteron 250mg injection per 3-4 weeks for 6 months
  Other Names: Sustanon 250mg

SUMMARY:
The study is designed to answer the following questions:

1. Is hypogonadism a cause for the metabolic syndrome ?
2. What is the effect of testosterone replacement on the metabolic parameters ?

DETAILED DESCRIPTION:
This is a retrospective design, which is performed by investigating the registrations of patients with hypogonadotrophic hypogonadism between the years 2002-2009.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Congenital hypogonadism
* Treatment Naive

Exclusion Criteria:

* Previous history of androgen replacement
* Hypertension
* Diabetes mellitus

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Mulligan T, Frick MF, Zuraw QC, Stemhagen A, McWhirter C. Prevalence of hypogonadism in males aged at least 45 years: the HIM study. Int J Clin Pract. 2006 Jul;60(7):762-9. doi: 10.1111/j.1742-1241.2006.00992.x. PMID 16846397
- [Background] Araujo AB, O'Donnell AB, Brambilla DJ, Simpson WB, Longcope C, Matsumoto AM, McKinlay JB. Prevalence and incidence of androgen deficiency in middle-aged and older men: estimates from the Massachusetts Male Aging Study. J Clin Endocrinol Metab. 2004 Dec;89(12):5920-6. doi: 10.1210/jc.2003-031719. PMID 15579737
- [Background] Saad F, Gooren LJ, Haider A, Yassin A. A dose-response study of testosterone on sexual dysfunction and features of the metabolic syndrome using testosterone gel and parenteral testosterone undecanoate. J Androl. 2008 Jan-Feb;29(1):102-5. doi: 10.2164/jandrol.107.002774. Epub 2007 Oct 3. PMID 17916569
- [Background] Koesling D, Schultz G, Bohme E. Sequence homologies between guanylyl cyclases and structural analogies to other signal-transducing proteins. FEBS Lett. 1991 Mar 25;280(2):301-6. doi: 10.1016/0014-5793(91)80317-v. PMID 1672855